CLINICAL TRIAL: NCT01229384
Title: Randomized Controlled Trial Comparing Standard Versus Positive Pressure Nebulization in Infants With Bronchiolitis to Reduce Hospital Admissions
Acronym: BPAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no enrollments, Trial administratively closed and withdrawn
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Principal Investigator, Mark Hostetler, Principal Investigator, Phoenix Children's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BronchPAP
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Bronchiolitis
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Positive Airway Pressure Nebulization (Experimental): Will administer nebulized medications using Positive Airway Pressure Nebulization
  Interventions: Device: Positive Airway Pressure nebulization
- Standard Nebulization (Active Comparator): Current standard of administering nebulized medications without positive airway pressure
  Interventions: Device: Standard passive nebulization of respiratory medications

INTERVENTIONS:
Device: Positive Airway Pressure nebulization — Using a device approved in pediatrics to deliver nebulized treatments of albuterol and racemic epinephrine with positive pressure
  Arms: Positive Airway Pressure Nebulization
Device: Standard passive nebulization of respiratory medications — Patients will receive standard passively inhaled nebulized albuterol and racemic epinephrine.
  Arms: Standard Nebulization

SUMMARY:
Hypothesis: That administration of nebulized therapy for bronchiolitis when using positive airway pressure is superior to standard mask ventilation in reducing hospital admissions.

Bronchiolitis is a lower respiratory tract infection (LRTI) syndrome caused by a variety of different viruses. It is the most common LRTI in children under 24 months old. Multiple studies have documented variation in treatment, hospitalization rates, and length of hospital stay for bronchiolitis, suggesting a lack of consensus and an opportunity to improve care for this common disorder.

Research to determine optimal delivery methods of respiratory medications that may augment oxygenation by decreasing atelectasis (Lung cell collapse) and increasing oxygen saturation have not been done. Currently bronchodilators are delivered through a passive process, inhaled as they are nebulized (made from liquid into gas) into a face mask. This study will evaluate whether using a newly developed positive pressure nebulization device that uses pressure to expand lung cells and, hypothetically, deliver the medication better, improves oxygenation by reducing atelectasis (lung cell collapse) to decrease hospitalization in infants with moderate to severe bronchiolitis.

Positive pressure nebulization is a relatively new adaptation of a previously existing modality, and is already currently in use here at PCH.

ELIGIBILITY:
Inclusion Criteria:

* Infants 2-24 months with moderate to severe bronchiolitis

Exclusion Criteria:

* Those outside the age range of 2-24 months, or less than postconceptual age of 48weeks for premature infants
* Those with comorbid conditions such as cyanotic heart disease, home oxygen use, tracheostomy use, or other serious medical conditions.
* Those with history of apnea

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Hospitalization Rates | 2 weeks
  Will measure rate of hospitalization of children comparing those treated with positive airway pressure nebulization and those with standard nebulization.

SECONDARY OUTCOMES:
Change in bronchiolitis Score | day of presentation
  Will measure change in bronchiolitis score by repiratory therapy of children comparing those treated with positive airway pressure nebulization and those with standard nebulization.
Change in Oxygen Saturation | Day of presentation
  Will measure change in oxygen saturation of children comparing those treated with positive airway pressure nebulization and those with standard nebulization.
Intensive Care Unit Admission Rate | day of presentation
  Will measure rate of hospitalization in the intensive care unit of children comparing those treated with positive airway pressure nebulization and those with standard nebulization.
Length of Stay | To be determined
  Will measure length of hospitalization of children comparing those treated with positive airway pressure nebulization and those with standard nebulization.
Unscheduled Return to the Emergency Department | 2 weeks
  Will measure rate of unscheduled return to the ED of children comparing those treated with positive airway pressure nebulization and those with standard nebulization.

CONTACTS AND LOCATIONS:
Overall Officials: Zebulon J Timmons, MD, Principal Investigator — Phoenix Children's Hospital; Mark Hostetler, MD, Study Director — Phoenix Children's Hospital

IPD SHARING:
Plan to Share IPD: Undecided